CLINICAL TRIAL: NCT03660904
Title: A Comparison Between Home-made Vitrification & Thawing Media and a Commercially Available Brand on Blastocyst Survival, Expansion and Implantation
Brief Title: A Comparison Between Home-made Vitrification & Thawing Media and a Commercially Available Brand on Blastocyst
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Saad, Assistant professor of Ob. & Gyn., Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Hawaa-3
Record Dates: First submitted 2018-09-02; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Blastocyst Disintegration
Keywords: vitrification; blastocysts; home-made media
MeSH Terms: conditions — Embryo Loss

STUDY DESIGN:
Intervention Model Description: Group 1 blastocysts were vitrified with the Vit (home made) HM according to shady grove protocol using open system on cryotop vit. device and thawed with gradual thawing technique using HM thawing media according to Kuwayama protocol.
  Group 2 blastocysts were cryopreserved with the Global Fast Freeze Kit using open system on cryotop vit. device and thawed using Global fast thaw kit. Blastocysts were assessed immediately for survival, subsequently cultured for 6-8 h, assessed for survival and expansion, then transferred and the percentages of Positive hCG, clinical pregnancy, implantation, multiple pregnancy and abortion were recorded.
Who Masked: Care Provider, Investigator
Masking Description: only the investigator knew the procedure and the media provided for each case
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home made media (Experimental): home made vitrification & thawing kit
  Interventions: Biological: home made vitrification & thawing kit
- Commercial media (Active Comparator): commercially available vitrification & thawing kit
  Interventions: Biological: commercially made vitrification & thawing kit

INTERVENTIONS:
Biological: home made vitrification & thawing kit — home made vitrification was made and prepared for vitrification of blastocysts then thawing with a prepared thawed media too
  Arms: Home made media
Biological: commercially made vitrification & thawing kit — commercially available vitrification & thawing kit were made and prepared for vitrification of blastocysts then thawing with a prepared thawed media too
  Arms: Commercial media

SUMMARY:
This study was conducted to evaluate and compare cryo-survival, re-expansion, and implantation rates of Day 5/6 human blastocysts that were vitrified with home-made media (HM) according to (Shady grove protocol) and warmed with gradual Thawing HM according to (Kuwayama protocol)with Global Fast Freeze/Thaw Kits (LifeGlobal, Canada).

DETAILED DESCRIPTION:
Group 1 blastocysts were vitrified with the Vit HM according to shady grove protocol using open system on cryotopvit. device and thawed with gradual thawing technique using HM according to Kuwayama protocol. Group 2 blastocysts were cryopreserved with the Global Fast Freeze Kitusing open system on cryotopvit. device and thawed using Gobal fast thaw kit. Blastocysts were subsequently cultured for 6-8 h, assessed for survival and expansion, then transferred and the percentages of Positive hCG, clinical pregnancy, implantation, multiple pregnancy and abortion were recorded.

ELIGIBILITY:
Inclusion Criteria:

* age of the patients 22-37
* All vitrified & thawed blastocyst.
* unexplained cases or ovarian factors for infertility.

Exclusion Criteria:

* extremes of age
* cases of uterine factor
* endometriosis

Ages: 22 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — blastocysts of infertile couples
Enrollment: 74 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
blastocyst immediate survival | 0 hour at time of thawing
  The effect of Vitrification protocol on the blastocyst immediate survival

SECONDARY OUTCOMES:
pregnancy rate | 2 weeks after transfer
  clinical pregnancy rate in these cases
live birth rate | 9 months
  live birth rate of positive pregnancy cases
Blastocyst survival at 6 hours | 6 hours after thawing
  The effect of Vitrification protocol on the blastocyst survival after 6 hours